CLINICAL TRIAL: NCT05568979
Title: Enhanced Passive Safety Surveillance of VaxigripTetra® (Quadrivalent Inactivated Split Virion Influenza Vaccine, Intramuscular Route) and Efluelda® (High-dose Quadrivalent Inactivated Split Virion Influenza Vaccine, Intramuscular Route) Vaccines in Europe During the Influenza Season 2022/23.
Brief Title: Safety Surveillance of VaxigripTetra® and Efluelda® Influenza Vaccines in Europe During the Influenza Season 2022/23
Status: Completed | Type: Observational
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: FLU00171; U1111-1271-1492 (Registry Identifier: ICTRP); FLU00171 (Other: Sanofi Identifier)
Record Dates: First submitted 2022-10-03; First posted 2022-10-06 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Influenza (Healthy Volunteers)
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- VaxigripTetra®: Participant vaccinated with VaxigripTetra® as per routine clinical practice
  Interventions: Biological: Quadrivalent Influenza Vaccine
- Efluelda®: Participant vaccinated with Efluelda® as per routine clinical practice
  Interventions: Biological: High-Dose Quadrivalent Influenza Vaccine

INTERVENTIONS:
Biological: Quadrivalent Influenza Vaccine — Intramuscular or subcutaneous administration
  Other Names: VaxigripTetra®
  Groups: VaxigripTetra®
Biological: High-Dose Quadrivalent Influenza Vaccine — Intramuscular administration
  Other Names: Efluelda®
  Groups: Efluelda®

SUMMARY:
This is an enhanced passive safety surveillance conducted in routine clinical care setting. Spontaneously reported ADRs will be collected by study staff following routine vaccination.

The primary objective of this surveillance is to estimate the vaccinee reporting rate (RR) of suspected adverse drug reactions (ADRs) occurring within 7 days following routine vaccination with VaxigripTetra® and Efluelda®, respectively, during the Northern Hemisphere (NH) influenza season 2022/23.

The secondary objectives of the study are:

* To estimate the vaccinee reporting rate of suspected ADRs occurring within 7 days following routine vaccination with VaxigripTetra® and Efluelda®, respectively, according to the pre-defined age groups (not applicable for Efluelda®)
* To estimate the vaccinee reporting rate of serious suspected ADRs after vaccination with VaxigripTetra® and Efluelda®, respectively, at any time following vaccination, within the EPSS

DETAILED DESCRIPTION:
Study duration per participant 2 months (including 6 weeks for VC distribution + 2 weeks for vaccinee reporting) following the first vaccination

ELIGIBILITY:
Inclusion Criteria:

* There are no formal inclusion criteria. Individuals who approach the site for vaccination and agree to receive a vaccination card will be included and vaccinated with the respective vaccine brand according to the country of their location,
* recommendations for the individual vaccines as well as national recommendations

Exclusion Criteria:

* none

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: VaxigripTetra® will be given to adults (including pregnant women) and children aged 6 months and older in Finland. Efluelda® will be given to adults 60 years of age and older in Germany.
Sampling Method: Non-Probability Sample
Enrollment: 1001 (Actual)
Dates: Start 2022-10-06 (Actual); Primary Completion 2022-11-29 (Actual); Study Completion 2022-11-29 (Actual)

PRIMARY OUTCOMES:
Vaccinee reporting rate of suspected adverse drug reactions (ADRs) following routine vaccination with VaxigripTetra® and Efluelda® | Within 7 days after vaccination
  Number of vaccinees who reported at least 1 suspected ADR divided by the total number of vaccination cards (VCs) distributed

SECONDARY OUTCOMES:
Vaccinees' reporting rate of ADRs according to age group | Within 7 days after vaccination
Vaccinees' reporting rate of serious suspected ADRs at any time following vaccination within the EPSS period | From vaccination to end of data collection (maximum 2 months following first vaccination)
  Serious suspected ADRs will be collected from vaccination up to the end of data collection. Data collection ends when 1000 vaccination cards have been distributed (per vaccine brand) plus 2 weeks or 2 months following the first vaccination, whichever comes first.
Vaccinees' reporting rate of suspected ADR at any time following vaccination within the EPSS period | From vaccination to end of data collection (maximum 2 months following first vaccination
  Suspected ADRs will be collected from vaccination up to the end of data collection. Data collection ends when 1000 vaccination cards have been distributed (per vaccine brand) plus 2 weeks or 2 months following the first vaccination, whichever comes first

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (15):
- Finland (6):
  - Investigational Site Number : 2-2-002, Helsinki
  - Investigational Site Number : 2-2-005, Jyväskylä
  - Investigational Site Number : 2-2-004, Kuopio
  - Investigational Site Number : 2-2-006, Rauma
  - Investigational Site Number : 2-2-003, Tampere
  - Investigational Site Number : 2-2-001, Turku
- Germany (9):
  - Investigational Site Number : 2760011, Berlin
  - Investigational Site Number : 2760005, Blankenhain
  - Investigational Site Number : 2760001, Donaueschingen
  - Investigational Site Number : 2760004, Düsseldorf
  - Investigational Site Number : 2760007, Frankfurt am Main
  - Investigational Site Number : 2760002, Fulda
  - Investigational Site Number : 2760003, Grafenrheinfeld
  - Investigational Site Number : 2760009, Martinsried
  - Investigational Site Number : 2760008, Wendelstein

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Result] Machado MAA, Gandhi-Banga S, Gallo S, Cousseau TG, Byrareddy RM, Nissila M, Schelling J, Monfredo C. Enhanced passive safety surveillance of high-dose and standard-dose quadrivalent inactivated split-virion influenza vaccines in Germany and Finland during the 2022/23 influenza season. Hum Vaccin Immunother. 2024 Dec 31;20(1):2322196. doi: 10.1080/21645515.2024.2322196. Epub 2024 Mar 6. PMID 38448394